CLINICAL TRIAL: NCT02902055
Title: Life-threatening Acute Respiratory Failure in Children: to Breathe or Not to Breathe Spontaneously, That's the Question
Brief Title: Paediatric Ards Neuromuscular Blockade Study
Acronym: PAN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19, slow enrolment
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Martin Kneyber, Chief, division of paediatric critical care medicine / Project leader, University Medical Center Groningen
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAN.1
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2024-01

CONDITIONS: ARDS
MeSH Terms: interventions — Neuromuscular Blocking Agents; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rocuronium 1 mg/kg i.v. (Active Comparator): Neuromuscular blocking agent
  Interventions: Drug: Neuromuscular Blocking Agents
- Isotonic saline (Active Comparator)
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Neuromuscular Blocking Agents — Neuromuscular blockae
  Arms: Rocuronium 1 mg/kg i.v.
Drug: Isotonic saline — Placebo
  Arms: Isotonic saline

SUMMARY:
Paediatric acute respiratory distress syndrome (ARDS) is a manifestation of severe, life-threatening lung injury. Care for paediatric patient is mainly supportive and based on what works in adults and personal experiences, including the use of mechanical ventilation. However, differences in lung physiology and immunology between (young) children and adults suggests that adaptation of adult practices into paediatrics may not be justified. A study in adults with severe ARDS showed that early use of neuromuscular blocking agents (NMBA) improved 90-day survival and increased time off the ventilator without increasing muscle weakness. It is unknown if this is also true for paediatric ARDS

ELIGIBILITY:
Inclusion criteria

* Informed consent
* Age younger than 5 years
* Need for mechanical ventilation with tidal volume 5 - 8 mL/kg ideal bodyweight and PEEP equal to or greater than 5 cmH2O
* Early moderate - to - severe paediatric acute respiratory distress syndrome originating from any cause, i.e. acute onset of disease, and oxygenation index greater than 12, and one or more (bilateral) infiltrates on chest radiograph, and no evidence of left ventricular failure or fluid overload, and within the first 48 hours of PICU admission
* Sedation defined by Comfort - B scale between 9 - 12

Exclusion criteria

* No informed consent
* Known allergy or intolerance to rocuronium
* Continuous administration of neuromuscular blockade prior at the time of meeting the criteria for PARDS
* Chronic respiratory failure on home ventilation
* Intracranial hypertension
* Bone marrow transplantation
* Immunocompromised patients (congenital or acquired)
* Pre-existing pulmonary hypertension
* Congenital heart disease with left - to - right shunting
* Cyanotic congenital heart disease
* Expected duration of mechanical ventilation less than 48 hours
* Withdrawal of life - sustaining treatment

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
the cumulative respiratory morbidity score 12 months after PICU discharge, adjusted for confounding by age, gestational age, family history of asthma and/or allergy, season in which questionnaire was filled out and parental smoking | 12 months after PICU discharge

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Rudolph MW, Slager S, Burgerhof JGM, van Woensel JBM, Alffenaar JC, Wosten-van Asperen RM, de Hoog M, IJland MM, Kneyber MCJ; SKIC research consortium. Paediatric Acute Respiratory Distress Syndrome Neuromuscular Blockade study (PAN-study): a phase IV randomised controlled trial of early neuromuscular blockade in moderate-to-severe paediatric acute respiratory distress syndrome. Trials. 2022 Jan 31;23(1):96. doi: 10.1186/s13063-021-05927-w. PMID 35101098